CLINICAL TRIAL: NCT00678028
Title: Association Between Deficiency of MBL (Mannose-Binding Lectin) and Polymorphisms in MBL2 Gene to Urinary Tract Infection
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Orna Nitzan, Ha'emek Medical Center, Afula, Israel
Other Study IDs: 0080-07-EMC
Record Dates: First submitted 2008-02-17; First posted 2008-05-15 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Recurrent Urinary Tract Infections
Keywords: MBL, UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood for genetic test and serum for MBL test
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to genetic polymorphism about 15%-30% of the world population have low levels of MBL (Mannose Binding Lectin) in serum (below 500ng/mL). Different studies reported correlation between polymorphism in the MBL gene with low levels of MBL in serum and higher frequency of recurrent infections, severity of sepsis, ARDS and other infections. Urinary Tract Infection (UTI) is one of the very common infection in women. Since MBL is part of the innate immunity and there are proofs of relation between patients with recurrent infections and lack of MBL, we decided to explore a possible relation between low levels of MBL and different genotypes of MBL in young women and the risk to develop recurrent UTI.

ELIGIBILITY:
Inclusion Criteria:

* women above 18 years old.
* premenopausal
* recurrent UTI

Exclusion Criteria:

* pregnancy
* immunocompromised
* active malignancy
* HIV carrier

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young women with recurrent UTI - study group and young women witout recurrent UTI - a control group
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Locations (1):
- Ha'Emek Medical Center, Afula, Israel